CLINICAL TRIAL: NCT02453191
Title: Neoadjuvant Intralesional Injection of Talimogene Laherparepvec With Concurrent Preoperative Radiation in Patients With Locally Advanced Soft Tissue Sarcomas
Brief Title: TVEC and Preop Radiation for Sarcoma (4 ml Dose)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Mohammed Milhem, Clinical Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201504731 (4 milliliter dose)
Record Dates: First submitted 2015-04-28; First posted 2015-05-25 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — talimogene laherparepvec; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Talimogene Laherparepvec in combination with radiotherapy
  Talimogene Laherparepvec Dose Levels:
  • Initial dose for all = talimogene laherparepvec up to 4.0 mL of 106 PFU/mL
  Interventions: Drug: Talimogene Laherparepvec; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Talimogene Laherparepvec
Radiation: Radiotherapy — Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of talimogene laherparepvec when combined with radiation therapy.

Approximately 30 people will take part in this study conducted by investigators at the University of Iowa.

DETAILED DESCRIPTION:
This is a single-arm open-label phase Ib and phase II clinical study assessing the safety and relative efficacy of concurrent talimogene laherparepvec in combination with radiotherapy in patients with soft tissue sarcomas. Patients will be treated with neoadjuvant radiation and weekly intratumoral injections of talimogene laherparepvec. Weekly injections of talimogene laherparepvec will be continued until surgery. Surgery will be performed 4-6 weeks from the end of radiation therapy to allow for resolution of acute toxicities per current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Histologically confirmed diagnosis of locally advanced STS that is unresectable with clear wide margins, for which preoperative radiotherapy is considered appropriate.

EXAMPLES:

* Resectable stage IIB, III, and IV disease that are not suitable for surgically resection alone due to inability to achieve clear margins.
* Including metastatic (stage IV) disease for which radiotherapy and surgical resection are indicated.
* Except certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, and bone sarcomas.
* Previous treatment: prior systemic anti-cancer treatment consisting of chemotherapy, immunotherapy, or targeted therapy are allowed provided therapy completed at least 1 year prior to enrollment.
* No prior Talimogene laherparepvec or tumor vaccines allowed.
* No prior radiation to the same tumor bed allowed.

  * Age ≥18 years.
  * Both men and women of all races and ethnic groups are eligible for this trial.
  * ECOG performance status ≤1.
  * Patient must have measurable disease:
* Tumor size at least ≥ 5 cm in the longest diameter as measured by CT scan or MRI for which radiation is feasible.

  * Patient must have injectable disease (direct injection or ultrasound guided).

Exclusion Criteria:

* Certain histologic subtypes: GIST, Desmoid, Ewing sarcoma, Kaposi sarcoma, and bone sarcomas.
* History or evidence of sarcoma associated with immunodeficiency states (e.g.: Hereditary immune deficiency, HIV, organ transplant or leukemia).
* Subjects with retroperitoneal and visceral sarcoma.
* History or evidence of gastrointestinal inflammatory bowel disease (ulcerative colitis or Crohn's disease) or other symptomatic autoimmune disease including, inflammatory bowel disease, or history of any poorly controlled or severe systemic autoimmune disease (i.e., rheumatoid arthritis, systemic lupus erythematosus, scleroderma, type I diabetes, or autoimmune vasculitis).
* History of other malignancy within the past 3 years except treated with curative intent and no known active disease present and has not received chemotherapy for ≥ 1 year before enrollment/randomization and low risk for recurrence.
* History of prior or current autoimmune disease.
* History of prior or current splenectomy or splenic irradiation.
* Active herpetic skin lesions
* Require intermittent or chronic treatment with an anti-herpetic drug (e.g., acyclovir), other than intermittent topical use.
* Any non-oncology vaccine therapies used for the prevention of infectious disease within 28 days prior to enrollment and during treatment period.
* Concomitant treatment with therapeutic anticoagulants such as warfarin.
* Known human immunodeficiency virus (HIV) disease (requires negative test for clinically suspected HIV infection).
* Acute or chronic hepatitis B or hepatitis C infection (requires negative test for clinically suspected hepatitis B or hepatitis C infection).
* Evidence of hepatitis B -

  1. Positive HBV surface antigen (indicative for chronic hepatitis B or recent acute hepatitis B).
  2. Negative HBV surface antigen but positive HBV total core antibody (indicative for resolved hepatitis B infection or occult hepatitis B) and detectable copies of HBV DNA by PCR (detectable HBV DNA copies suggest occult hepatitis B).
* Evidence of hepatitis C -

  1. Positive HCV antibody and positive HCV RNA by PCR (undetectable RNA copies suggest past and resolved hepatitis C infection).
* Female subjects who are pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of study treatment.
* Female subjects of childbearing potential or male subjects who are unwilling to use 2 highly effective methods of contraception during study treatment and through 3 months after the last dose of study treatment. See Section 7.5 for more details.
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
* Other investigational procedures while participating in this study that could affect the primary objective of the study as determined by the PI are excluded.
* Subject previously has entered this study.
* Patients who are receiving any other investigational agents.
* Evidence of CNS metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talimogene laherparepvec.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients on or requiring immunosuppressive therapies.
* Any of the following laboratory abnormalities:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count (ANC) < 1500 per mm3
  * Platelet count < 100,000 per mm3
  * Total bilirubin > 1.5 × ULN
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN
  * Alkaline phosphatase > 2.5 × ULN
  * PT (or INR) and PTT (or aPTT) > 1.5 × ULN
  * Creatinine > 2.0 × ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monga V, Miller BJ, Tanas M, Boukhar S, Allen B, Anderson C, Stephens L, Hartwig S, Varga S, Houtman J, Wang L, Zhang W, Jaber O, Thomason J, Kuehn D, Rajput M, Metz C, Zamba KD, Mott S, Abanonu C, Bhatia S, Milhem M. Intratumoral talimogene laherparepvec injection with concurrent preoperative radiation in patients with locally advanced soft-tissue sarcoma of the trunk and extremities: phase IB/II trial. J Immunother Cancer. 2021 Jul;9(7):e003119. doi: 10.1136/jitc-2021-003119. PMID 34330766

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: talimogene laherparepvec in combination with radiotherapy
  talimogene laherparepvec: talimogene laherparepvec
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Period: Overall Study
Arm/Group | Treatment
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 7 subjects enrolled in the Phase 1b portion, 23 subjects enrolled in the Phase 2 portion of the study
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 61 [28 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: A DLT is defined as any of the following talimogene laherparepvec-related toxicity or related to the combination of talimogene laherparepvec and radiation therapy during treatment and up to 4 weeks after the last talimogene laherparepvec injection: Grade 3 or greater immune-mediated adverse events, Grade 3 or greater allergic reactions, any grade plasmacytoma, any other unexpected grade 3 or greater hematologic or non-hematologic toxicity, with the exceptions of: any grade of alopecia, expected radiation related skin toxicity of any grade, Grade 3 arthralgia or myalgia, brief (< 1 week) grade 3 fatigue, Grade 3 fever, Grade 3 diarrhea or vomiting responding to supportive case.
Time Frame: 14 weeks
Population: 6 participants were evaluable for DLT assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Phase 2: Pathologic Tumor Necrosis Rate
Description: Pathologic tumor necrosis rate is defined as the percentage of subjects with pathologic tumor necrosis ≥ 95%.
Time Frame: 14 weeks
Population: In Phase 2, 24 subjects were accrued. One patient refused surgery resulting in 23 subjects being evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 23
Participants
  < 95% | 18
  ≥ 95% | 5

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of patients with a confirmed complete or partial response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI/CT:
  Complete response (CR) is the disappearance of all target lesions. Partial response (PR) is a 30% decrease in the sum of the longest dimensions of the target lesions, relative to baseline. Progressive disease (PD) is an increase of 20% or more in the sum of the longest dimension of target lesions. Stable disease (SD) is a decrease in the tumor size of < 30% or an increase of < 20%.
Time Frame: 24 months
Population: Subjects completing Phase 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 20
  Progressive Disease | 9

4. Secondary Outcome: Percentage of Participants With 2 Year Progression-Free Survival
Description: Progression-free survival is defined as the time from treatment initiation to the date of first documentation of disease progression or death due to any cause. Otherwise, patients are censored at the date of last radiographic assessment for progression.
Time Frame: 24 months
Population: Subjects completing Phase 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of participants | 57 [37 to 72]

5. Secondary Outcome: Percentage of Participants With 2 Year Overall Survival
Description: Overall survival is defined as the time from treatment initiation to death due to any cause. Patients still alive are censored at last date known to be alive.
Time Frame: 24 months
Population: Subjects in Phase 1 and 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment: Talimogene Laherparepvec in combination with radiotherapy
  Talimogene Laherparepvec Dose Levels:
  • Initial dose for all = talimogene laherparepvec up to 4.0 mL of 106 PFU/mL
  Talimogene Laherparepvec: Talimogene Laherparepvec
  Radiotherapy: Concurrent Preoperative Radiation. External Beam Radiation Therapy (EBRT) will be given at the standard dose for resectable soft tissue sarcomas. according to the NCCN sarcoma guidelines.
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of participants | 77 [57 to 88]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: To further assess the safety of talimogene laherparepvec given concurrently with preoperative external beam radiation in sarcoma patients.Information regarding the occurrence of adverse events will be collected from the time the subject signs the informed consent form and throughout their participation in the study, including a period of 30 days after the last dose of study drug.
Time Frame: 14 weeks
Population: All 30 enrolled subjects were assessed for AEs
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: Information regarding the occurrence of adverse events was collected from the time the subject signed the informed consent form and throughout their participation in the study, through a period of 30 days after the last dose of study drug, up to 14 weeks.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Flushing (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (19)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6)
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 6 (8)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, (Renal and urinary disorders) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 5 (13)
Delirium (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (2)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (15)
Dysgeusia (Nervous system disorders) | 5 (8)
Headache (Nervous system disorders) | 15 (26)
Nervous system disorders - Other, (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Tremor (Nervous system disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (22)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (16)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 8 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Alanine aminotransferase (Investigations) | 6 (8)
Alkaline phosphatase increased (Investigations) | 4 (5)
Carbon monoxide diffusing capacity (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (8)
Lymphocyte count decreased (Investigations) | 10 (30)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 4 (4)
Weight loss (Investigations) | 6 (11)
White blood cell decreased (Investigations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 26 (63)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural (Injury, poisoning and procedural complications) | 2 (4)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Infections and infestations - Other, (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 2 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Immune system disorders - Other, (Immune system disorders) | 1 (1)
Chills (General disorders) | 18 (46)
Edema limbs (General disorders) | 12 (19)
Fatigue (General disorders) | 26 (71)
Fever (General disorders) | 12 (16)
Flu like symptoms (General disorders) | 14 (48)
General disorders and administration site (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Injection site reaction (General disorders) | 5 (10)
Localized edema (General disorders) | 3 (5)
Malaise (General disorders) | 4 (7)
Non-cardiac chest pain (General disorders) | 1 (3)
Pain (General disorders) | 18 (52)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (14)
Diarrhea (Gastrointestinal disorders) | 9 (24)
Dry mouth (Gastrointestinal disorders) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (39)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (28)
Eye disorders - Other, specify (Eye disorders) | 1 (2)
Photophobia (Eye disorders) | 1 (5)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (9)
Vertigo (Ear and labyrinth disorders) | 2 (7)
Heart failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 4 (8)
Anemia (Blood and lymphatic system disorders) | 21 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT02453191/Prot_SAP_002.pdf
  • Informed Consent Form (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02453191/ICF_003.pdf